CLINICAL TRIAL: NCT00835965
Title: A Randomized, Double-Blind Comparison of Oral Aprepitant and Lower Dose Dexamethasone vs Aprepitant Alone for Preventing Postoperative Nausea and Vomiting After Elective Laparoscopic Surgeries
Brief Title: Oral Aprepitant and Lower Dose Dexamethasone Versus Aprepitant Alone for Preventing Postoperative Nausea and Vomiting (PONV) After Elective Laparoscopic Surgeries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Main Line Health (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Drexel University College of Medicine (Other)
Responsible Party: Dmitri Chamchad, MD, Main Line Health System, Lankenau Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Merck-Chamchad-2008; Merck #32589
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Last update posted 2009-02-04 (Estimated); Status verified 2009-02

CONDITIONS: Nausea; Vomiting
Keywords: Laparoscopic; Surgery; Postoperative; Nausea; Vomiting; Aprepitant; Dexamethasone; Postoperative Nausea, Postoperative Vomiting
MeSH Terms: conditions — Nausea; Vomiting; Postoperative Nausea and Vomiting | interventions — Dexamethasone; Aprepitant

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Comparator (Active Comparator): Patients receive aprepitant and dexamethasone for prevention of postoperative nausea and vomiting
  Interventions: Drug: Dexamethasone; Drug: Aprepitant
- Placebo Comparator (Placebo Comparator): Patients receiving aprepitant and placebo dexamethasone for prevention of postoperative nausea and vomiting
  Interventions: Drug: Aprepitant; Drug: Placebo Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone 5 mg administered intravenously following endotracheal intubation
  Other Names: EMEND
  Arms: Active Comparator
Drug: Aprepitant — Aprepitant 40mg PO one time at least one hour prior to induction of anesthesia
  Other Names: EMEND
Drug: Placebo Dexamethasone
  Arms: Placebo Comparator

SUMMARY:
The combination of aprepitant and lower dose dexamethasone is superior to aprepitant alone with respect to the proportion of patients with a complete response (no vomiting and no use of rescue therapy) during 24 hours after the placement of last suture/staple.

DETAILED DESCRIPTION:
Postoperative Nausea and Vomiting (PONV) is a serious and common (50%-70%) complication of laparoscopic abdominal surgery. PONV is multifactorial, and the treatment is multimodal. Preoperative treatment should target the specific mechanism of PONV to minimize its incidence/consequences to the benefit of the patients.

Aprepitant, a selective antagonist of neurokinin-1 (NK-1) receptors, blocks the emetic effects of substance P.5 Substance P action on the NK-1 receptors in the central nervous system (CNS) is one of the final pathways to an emetic response. Dexamethasone is an inexpensive and effective antiemetic drug with minimal side effects after a single-dose administration. The commonly used minimal effective dose is 8 to 10 mg, but the dose 5 mg is suggested for PONV in patients undergoing laparoscopic surgeries. Based on the literature review, occurrence of PONV does not significantly differ at dosing of Dexamethasone equal or higher than 4 mg.

This study compares the incidence of nausea, vomiting, need for rescue medication, prolonged PACU time, and unplanned hospital admission in patients with high risk for PONV treated with oral aprepitant and dexamethasone or aprepitant alone preoperatively.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* ASA physical status I-III
* must have at least 2 risk factors for PONV

Exclusion Criteria:

* pregnant or breast feeding patients
* antiemetic medication in previous 24 hours
* allergy or other contraindication to study medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-02; Primary Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
the incidences of nausea, vomiting, need for rescue medication | 1 hour, 2 hours, 24 hours after surgery

SECONDARY OUTCOMES:
incidences of unplanned hospital admission; duration of PACU stay | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Dmitri Chamchad, MD, Principal Investigator — Lankenau Hospital, Lankenau Institute for Medical Research
Locations (1):
- Lankenau Hospital, Wynnewood, Pennsylvania, United States